CLINICAL TRIAL: NCT00914329
Title: Randomized Controlled Study Versus Placebo Evaluating Effectiveness of Gelsemium Sempervirens (5CH et 15CH) on Provoked Anticipatory Anxiety, in Healthy Volunteers
Brief Title: Gelsemium Sempervirens in Anticipatory Anxiety
Acronym: ANXIHOMEV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: BOIRON (Industry)
Responsible Party: Mr FrédérickMarie, CHU de Grenoble
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCIC 08 20
Record Dates: First submitted 2009-05-29; First posted 2009-06-05 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Anxiety
Keywords: stress provoked; healthy volunteers; gelsemium; homeopathy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gelsemium 5CH (Experimental): Globules of Gelsemium sempervirens 5CH
  Interventions: Drug: Gelsemium Sempervirens
- Gelsemium 15CH (Experimental): Globules of Gelsemium Sempervirens 15CH
  Interventions: Drug: Gelsemium Sempervirens
- Placebo (Placebo Comparator): Globules of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gelsemium Sempervirens — 5CH, one dose of globules morning and evening during 2 days plus one dose the morning of the day of the stress-test.
  Arms: Gelsemium 5CH
Drug: Gelsemium Sempervirens — 15CH, one dose of globules morning and evening during 2 days plus one dose the morning of the day of the stress-test.
  Arms: Gelsemium 15CH
Drug: Placebo — placebo, one dose of globules morning and evening during 2 days plus one dose the morning of the day of the stress-test.
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of Gelsemium sempervirens 5CH et 15CH on anticipatory provoked anxiety, in healthy volunteers.

DETAILED DESCRIPTION:
State-anxiety can appear during banal events without objective harrowing factors. It is preponderant in particular situations as exams and competitive examination for example, and may be responsible of failures, notably at school. Particularly, a form of anxiety said anticipatory (largely named nerves) is focused on a coming performance. This anticipative anxiety, maximal before the beginning of the test, disappears during this test to let place to relief. Even if phenomenon of habituation exists, it can be responsible of social and professional failures.

Numerous therapeutics exists to fight against anxiety, non medicinal first but the resort to drugs are sometime necessary. The reference is the class of benzodiazepines. Many patients try non conventional medicines, like homeopathy.

Gelsemium sempervirens would be active on sensible et emotional persons, reducing anxiety in some situations. A large used of Gelsemium sempervirens is the case of a situation of provoked stress in particular exam. That is the reason why the drug is particularly intended to a population of young adults who don't want to use " traditional " tranquillizing. But this drug, largely used, has never showed his effectiveness on provoked anxiety, in biomedical research. That is why we proposed in this study to compare the effectiveness of Gelsemium sempervirens 5CH, Gelsemium sempervirens 15CH and placebo, in a situation of provoked anxiety in young adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman,
* age between 18 et 40 ans,
* affiliated to a regime of social security or equivalent

Exclusion Criteria:

* Medical history of psychiatric disease relevant of psychoses,
* Medical history of hospitalisation in psychiatric environment,
* psychotropic substance of the class of antidepressants, antipsychotics and normothymics), in the year before inclusion,
* Taking, even punctual of psychotropics substances of the class of benzodiazepines and related, in the month before inclusion,
* Taking, even punctual of psychotropics substances of the class of anxiolytics non benzodiazepines, in the month before inclusion: meprobamate, hydroxyzine, buspirone, captodiamine, pregabalin, etifoxine,
* Taking, even punctual of substances of the class of the sedatives divers, in the month before inclusion: phytotherapy, homeopathy, sedatives with brome, mineral elements,
* Taking, even punctual of substances of the class of antihistamine with hypnotic aim, in the month before inclusion,
* Taking, even punctual of propanolol in the month before inclusion
* Known Addiction,
* Handicap incompatible with the Stress Test : blindness, partially sighted, daltonism, dementia, language troubles,
* Pregnancy, parturient and nursing woman,
* Person private of freedom by judicial or administrative decision, person under measure of legal protection,
* allergy to one of the constituents

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Anxiety level evaluated by the STAI-E, in absolute value and et difference with basal state, according to the treatment received by the volunteers (Gelsemium sempervirens 5CH, 15CH or placebo) | day 0

SECONDARY OUTCOMES:
anxiety level measured by the visual analogic scale of anxiety, in absolute value and difference with the basal state, according to the treatment received by the volunteers (Gelsemium sempervirens 5CH, 15CH or placebo) | day -7, day -5 and day 0
anxiety level measured by the scale of anxiety state in competition (EEAC), in absolute value and difference with the basal state, according to the treatment received by the volunteers (Gelsemium sempervirens 5CH, 15CH or placebo) | day 0
Continue measure of arterial pressure, heart rate, respiratory rate, according to the treatment received by the volunteers (Gelsemium sempervirens 5CH, 15CH or placebo) | day 0
anxiety measured by STAI-T | day -7 and day -5
score of stress-test | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD, PhD, Principal Investigator — CIC, CHU Grenoble
Locations (1):
- Clinical Research Center, Grenoble, France

REFERENCES:
- [Background] Binsard AM, Guillemain J, Platel A, Savini EC, Tetau M. Etude psychopharmacologique de dilution homéopathiques de Gelsemium et d'Ignatia. Ann Homeop Fr. 22: 35-50; 1980.
- [Background] Nasolotsiry E. Raveloson ; R. Rasoloherimampiononiaina ; A. Ramialiharisoa. Indication homéopathique en prémédication anesthésique. Correspondance homéoweb.